CLINICAL TRIAL: NCT05141162
Title: The Effect of Knitting on Mothers' Anxiety Levels During Pediatric Hernia Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Güzide Özden AKCAN, Student, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: anxiety and knitting
Record Dates: First submitted 2021-01-14; First posted 2021-12-02 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Mothers
Keywords: Knitting; anxiety; hernia; art therapy
MeSH Terms: conditions — Anxiety Disorders; Hernia | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- case group (Experimental): In the first stage, an information form including socio-demographic characteristics prepared within the framework of the literature and State-Trait Anxiety Inventory will be applied to mothers before surgery. Later, the experimental group will be knitted by the researcher during the surgical operation. The necessary materials (knitting needle and thread) for the knitting attempt will be given to the participants in the experimental group by the researcher. A neutral color, white, will be used as the knitting yarn color. Knitting will start 15 minutes after the child enters the operation and will be knitted for 30-40 minutes on average. At the end of the surgery, the State-Trait Anxiety Inventory scale will be applied again to evaluate the anxiety levels of the participants in the experimental and control groups. The vital signs of the mothers will be measured at the beginning of the operation and close to the end of the operation.
  Interventions: Behavioral: case and control group
- control group (No Intervention): An information form including socio-demographic characteristics prepared within the framework of the preoperative literature and State-Trait Anxiety Inventory will be applied to mothers. No attempt will be made to this group. At the end of the surgery, the State Trait Anxiety Inventory scale will be applied again to evaluate the anxiety levels of the participants in the experimental and control groups. The vital signs of the mothers will be measured at the beginning of the operation and near the end of the operation.

INTERVENTIONS:
Behavioral: case and control group — randomized controlled experimental study
  Arms: case group

SUMMARY:
Regardless of the type of surgical intervention, it is a negative life experience for the child and family members and is known to cause anxiety. Having a surgical incision in the child's body and the likelihood of developing conditions such as pain, organ loss or death, change in the parental role, and the hospital environment are situations that increase the stress of the parents. Hernia is the most common surgical pathology in children. Hernias are also risky in terms of complications.

Parents' experiencing severe anxiety may prevent their ability to understand the child's explanations correctly, interpret events realistically, make correct decisions, participate in the care of the child, and use appropriate coping methods. Parents abandon their habitual attitudes because they feel anxiety and sadness. Their tolerance increases and, as a result, they do whatever their children want. This change in the attitudes of the parents may increase the anxiety of the child and make him feel more sick than he is. Therefore, it is very important for the child to reduce the parent's anxiety.

At the pathological level, anxiety requires pharmacological and / or psychosocial intervention. The main purpose of psychosocial intervention is to understand and discover one's emotions. Some authors mention the benefits of using expressive methods. Art practices are at the top of the expressionist methods, and according to the nursing interventions classification system (NIC), art therapy is among the nursing interventions.

DETAILED DESCRIPTION:
Studies have shown that art practices reduce women's stress, anxiety, depression and fatigue. On the other hand, occupational therapy is another example of the use of art in psychotherapy. Various crafts and decorations are made in this type of therapy.

Most of the studies on knitting in the literature have been conducted with groups, and there is no study examining the effect of knitting in reducing the anxiety of mothers whose children underwent surgery. In this study, which was planned as a randomized controlled experimental study, it was aimed to examine the effect of knitting on the anxiety levels of the mothers of children who underwent hernia surgery.

The objectives of the study; To determine the anxiety levels of mothers of children who underwent planned surgery. To determine the effects of demographic characteristics on mothers' anxiety levels. To determine the effect of knitting knitting method on the anxiety levels of the mothers of children who underwent hernia surgery.

ELIGIBILITY:
* Inclusion criteria in the study;

  1. Mothers know how to knit,
  2. Mothers' willingness to participate in the study,
  3. The child has not had a previous surgical operation.
  4. The mother has not had any psychological trauma or psychiatric diagnosis in the last six months.

exclusion criteria in the study;

1. Mothers do not know how to knit,
2. Refusal of mothers to participate in research,
3. The child has had previous surgery,
4. The mother's history of any psychological trauma or psychiatric diagnosis in the last six months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Research evidence shows that especially mothers have a high level of anxiety during surgery.
Enrollment: 90 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Anxiety Levels of Mothers | 15 minutes after the start of surgery
  Anxiety Levels of Mothers will be defined with the State-Trait Anxiety Inventory.
Anxiety Levels of Mothers | 1 hour after the start of surgery
  Anxiety Levels of Mothers will be defined with the State-Trait Anxiety Inventory.
Heartbeat of mothers | 15 minutes after the start of surgery
  heartbeat per minutes
Heartbeat of mothers | 1 hour after the start of surgery
  heartbeat per minutes
Breathing rate of mothers | 15 minutes after the start of surgery
  breathing rate per minutes
Breathing rate of mothers | 1 hour after the start of surgery
  breathing rate per minutes
Blood pressure of mothers | 15 minutes after the start of surgery
  blood pressure in mmHg
Blood pressure of mothers | 1 hour after the start of surgery
  blood pressure in mmHg
Oxygen saturation of mothers | 15 minutes after the start of surgery
  oxygen saturation in percent
Oxygen saturation of mothers | 1 hour after the start of surgery
  oxygen saturation in percent

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences Universyt, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar A, Das S, Chauhan S, Kiran U, Satapathy S. Perioperative Anxiety and Stress in Children Undergoing Congenital Cardiac Surgery and Their Parents: Effect of Brief Intervention-A Randomized Control Trial. J Cardiothorac Vasc Anesth. 2019 May;33(5):1244-1250. doi: 10.1053/j.jvca.2018.08.187. Epub 2018 Aug 22. PMID 30243867
- [Background] Pomicino L, Maccacari E, Buchini S. Levels of anxiety in parents in the 24 hr before and after their child's surgery: A descriptive study. J Clin Nurs. 2018 Jan;27(1-2):278-287. doi: 10.1111/jocn.13895. Epub 2017 Dec 11. PMID 28544343
- [Background] Brooks L, Ta KN, Townsend AF, Backman CL. "I just love it": Avid knitters describe health and well-being through occupation. Can J Occup Ther. 2019 Apr;86(2):114-124. doi: 10.1177/0008417419831401. Epub 2019 Mar 11. PMID 30857405
- [Background] Pollanen S. The meaning of craft: craft makers' descriptions of craft as an occupation. Scand J Occup Ther. 2013 May;20(3):217-27. doi: 10.3109/11038128.2012.725182. Epub 2012 Sep 19. PMID 22989300